CLINICAL TRIAL: NCT04640870
Title: An Observational Study to Assess the Molecular Epidemiology of Epidermal Growth Factor Receptor (EGFR) Mutations in Patients With Advanced EGFR Mutation-positive Non-small Cell Lung Cancer Treated With Afatinib in Real-world Clinical Set-tings in Greece
Brief Title: The Molecular Epidemiology of Epidermal Growth Factor Receptor (EGFR) Mutations in Patients With Advanced EGFR Mutation-positive Non-small Cell Lung Cancer Treated With Afatinib
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: ΗΕ2/15
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Non Small Cell Lung Cancer; EGF-R Positive Non-Small Cell Lung Cancer; EGFR Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Afatinib — Treatment with Afatinib, any line, in metastatic, EGFR mutated patients with NSCLC

SUMMARY:
This is an observational, non-interventional, single-country, multi center, retrospective cohort study, based on real world data collection, of patients with locally advanced or metastatic Epidermal Growth Factor Receptor (EGFR) mutation-positive Non-Small Cell Lung Cancer (NSCLC) who had been treated with Afatinib at any line.

DETAILED DESCRIPTION:
This is an observational, non-interventional, single-country, multicenter, retrospective cohort study, based on real world data collection, of patients with locally advanced or metastatic EGFR mutation-positive NSCLC who had been treated with Afatinib s at any line.

The study is carried out by hospital-based oncologists/pneumonologists specializing in lung cancer under real-world conditions of daily clinical practice. Investigators were selected through a documented and structured feasibility process which accounted for physicians' qualifications, previous participation and experience in similar clinical studies, recruitment potential, and retention capability. In addition, in order to represent variations in current real-world patterns of care, research sites were recruited from various geographic regions in Greece, also taking into consideration the regional setting and type of healthcare site/institution (publicly/privately owned, specialized oncology/pulmonology clinic, university clinic).

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Patients diagnosed with Non-small cell lung cancer
* metastatic disease
* Afatinib treated in any line
* EGFR mutated

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective analysis of patients with histologically confirmed Non-small cell lung cancer and EGFR mutated, with progressive disease. Patients analysed in this study have been treated with Afatinib in any line. Patients have been treated in Hellenic Cooperative Oncology Group(HeCOG)- affiliated departments of oncology.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | From Day 1 of treatment with Afatinib until disease progression, death from any cause or last follow-up, whichever occurs first, up to 12 months
  Progression Free Survival

SECONDARY OUTCOMES:
Overall survival | From Day 1 of treatment with Afatinib until death from any cause or last follow-up, up to 24 months
  Overall survival
Second progression-free survival (PFS2) | From the initiation of next treatment following discontinuation of Afatinib to the date of progression, death or last contact, up to 6 months
  Second progression-free survival (PFS2)
Assessment of the safety profile of Afatinib | In every cycle, every 28 days
  assessment of the safety profile of Afatinib

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Mountzios, MD, Principal Investigator — Henry Dunant Hospital Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Planchard D, Popat S, Kerr K, Novello S, Smit EF, Faivre-Finn C, Mok TS, Reck M, Van Schil PE, Hellmann MD, Peters S; ESMO Guidelines Committee. Metastatic non-small cell lung cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv192-iv237. doi: 10.1093/annonc/mdy275. No abstract available. PMID 30285222
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Background] Mitsudomi T, Morita S, Yatabe Y, Negoro S, Okamoto I, Tsurutani J, Seto T, Satouchi M, Tada H, Hirashima T, Asami K, Katakami N, Takada M, Yoshioka H, Shibata K, Kudoh S, Shimizu E, Saito H, Toyooka S, Nakagawa K, Fukuoka M; West Japan Oncology Group. Gefitinib versus cisplatin plus docetaxel in patients with non-small-cell lung cancer harbouring mutations of the epidermal growth factor receptor (WJTOG3405): an open label, randomised phase 3 trial. Lancet Oncol. 2010 Feb;11(2):121-8. doi: 10.1016/S1470-2045(09)70364-X. Epub 2009 Dec 18. PMID 20022809
- [Background] Inoue A, Kobayashi K, Maemondo M, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Updated overall survival results from a randomized phase III trial comparing gefitinib with carboplatin-paclitaxel for chemo-naive non-small cell lung cancer with sensitive EGFR gene mutations (NEJ002). Ann Oncol. 2013 Jan;24(1):54-9. doi: 10.1093/annonc/mds214. Epub 2012 Sep 11. PMID 22967997
- [Background] Wu YL, Zhou C, Hu CP, Feng J, Lu S, Huang Y, Li W, Hou M, Shi JH, Lee KY, Xu CR, Massey D, Kim M, Shi Y, Geater SL. Afatinib versus cisplatin plus gemcitabine for first-line treatment of Asian patients with advanced non-small-cell lung cancer harbouring EGFR mutations (LUX-Lung 6): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Feb;15(2):213-22. doi: 10.1016/S1470-2045(13)70604-1. Epub 2014 Jan 15. PMID 24439929
- [Background] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L; Spanish Lung Cancer Group in collaboration with Groupe Francais de Pneumo-Cancerologie and Associazione Italiana Oncologia Toracica. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2012 Mar;13(3):239-46. doi: 10.1016/S1470-2045(11)70393-X. Epub 2012 Jan 26. PMID 22285168
- [Background] Paz-Ares L, Tan EH, O'Byrne K, Zhang L, Hirsh V, Boyer M, Yang JC, Mok T, Lee KH, Lu S, Shi Y, Lee DH, Laskin J, Kim DW, Laurie SA, Kolbeck K, Fan J, Dodd N, Marten A, Park K. Afatinib versus gefitinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: overall survival data from the phase IIb LUX-Lung 7 trial. Ann Oncol. 2017 Feb 1;28(2):270-277. doi: 10.1093/annonc/mdw611. PMID 28426106
- [Background] Park K, Tan EH, O'Byrne K, Zhang L, Boyer M, Mok T, Hirsh V, Yang JC, Lee KH, Lu S, Shi Y, Kim SW, Laskin J, Kim DW, Arvis CD, Kolbeck K, Laurie SA, Tsai CM, Shahidi M, Kim M, Massey D, Zazulina V, Paz-Ares L. Afatinib versus gefitinib as first-line treatment of patients with EGFR mutation-positive non-small-cell lung cancer (LUX-Lung 7): a phase 2B, open-label, randomised controlled trial. Lancet Oncol. 2016 May;17(5):577-89. doi: 10.1016/S1470-2045(16)30033-X. Epub 2016 Apr 12. PMID 27083334
- [Background] Wu YL, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Tsuji F, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Nadanaciva S, Sandin R, Mok TS. Dacomitinib versus gefitinib as first-line treatment for patients with EGFR-mutation-positive non-small-cell lung cancer (ARCHER 1050): a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1454-1466. doi: 10.1016/S1470-2045(17)30608-3. Epub 2017 Sep 25. PMID 28958502
- [Background] Mok TS, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Lee M, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Wu YL. Improvement in Overall Survival in a Randomized Study That Compared Dacomitinib With Gefitinib in Patients With Advanced Non-Small-Cell Lung Cancer and EGFR-Activating Mutations. J Clin Oncol. 2018 Aug 1;36(22):2244-2250. doi: 10.1200/JCO.2018.78.7994. Epub 2018 Jun 4. PMID 29864379
- [Background] Wang J, Wang B, Chu H, Yao Y. Intrinsic resistance to EGFR tyrosine kinase inhibitors in advanced non-small-cell lung cancer with activating EGFR mutations. Onco Targets Ther. 2016 Jun 22;9:3711-26. doi: 10.2147/OTT.S106399. eCollection 2016. PMID 27382309
- [Background] Gainor JF, Shaw AT. Emerging paradigms in the development of resistance to tyrosine kinase inhibitors in lung cancer. J Clin Oncol. 2013 Nov 1;31(31):3987-96. doi: 10.1200/JCO.2012.45.2029. Epub 2013 Oct 7. PMID 24101047
- [Background] Kim HR, Cho BC, Shim HS, Lim SM, Kim SK, Chang J, Kim DJ, Kim JH. Prediction for response duration to epidermal growth factor receptor-tyrosine kinase inhibitors in EGFR mutated never smoker lung adenocarcinoma. Lung Cancer. 2014 Mar;83(3):374-82. doi: 10.1016/j.lungcan.2013.12.011. Epub 2014 Jan 3. PMID 24468202
- [Background] Levy BP, Rao P, Becker DJ, Becker K. Attacking a Moving Target: Understanding Resistance and Managing Progression in EGFR-Positive Lung Cancer Patients Treated With Tyrosine Kinase Inhibitors. Oncology (Williston Park). 2016 Jul;30(7):601-12. PMID 27432364
- [Background] Cortot AB, Janne PA. Molecular mechanisms of resistance in epidermal growth factor receptor-mutant lung adenocarcinomas. Eur Respir Rev. 2014 Sep;23(133):356-66. doi: 10.1183/09059180.00004614. PMID 25176972
- [Background] Yu HA, Arcila ME, Rekhtman N, Sima CS, Zakowski MF, Pao W, Kris MG, Miller VA, Ladanyi M, Riely GJ. Analysis of tumor specimens at the time of acquired resistance to EGFR-TKI therapy in 155 patients with EGFR-mutant lung cancers. Clin Cancer Res. 2013 Apr 15;19(8):2240-7. doi: 10.1158/1078-0432.CCR-12-2246. Epub 2013 Mar 7. PMID 23470965
- [Background] Blakely CM, Bivona TG. Resiliency of lung cancers to EGFR inhibitor treatment unveiled, offering opportunities to divide and conquer EGFR inhibitor resistance. Cancer Discov. 2012 Oct;2(10):872-5. doi: 10.1158/2159-8290.CD-12-0387. PMID 23071030
- [Background] Sequist LV, Waltman BA, Dias-Santagata D, Digumarthy S, Turke AB, Fidias P, Bergethon K, Shaw AT, Gettinger S, Cosper AK, Akhavanfard S, Heist RS, Temel J, Christensen JG, Wain JC, Lynch TJ, Vernovsky K, Mark EJ, Lanuti M, Iafrate AJ, Mino-Kenudson M, Engelman JA. Genotypic and histological evolution of lung cancers acquiring resistance to EGFR inhibitors. Sci Transl Med. 2011 Mar 23;3(75):75ra26. doi: 10.1126/scitranslmed.3002003. PMID 21430269
- [Background] Takeda M, Nakagawa K. First- and Second-Generation EGFR-TKIs Are All Replaced to Osimertinib in Chemo-Naive EGFR Mutation-Positive Non-Small Cell Lung Cancer? Int J Mol Sci. 2019 Jan 3;20(1):146. doi: 10.3390/ijms20010146. PMID 30609789
- [Background] Wu SG, Liu YN, Tsai MF, Chang YL, Yu CJ, Yang PC, Yang JC, Wen YF, Shih JY. The mechanism of acquired resistance to irreversible EGFR tyrosine kinase inhibitor-afatinib in lung adenocarcinoma patients. Oncotarget. 2016 Mar 15;7(11):12404-13. doi: 10.18632/oncotarget.7189. PMID 26862733
- [Background] Oxnard GR, Arcila ME, Sima CS, Riely GJ, Chmielecki J, Kris MG, Pao W, Ladanyi M, Miller VA. Acquired resistance to EGFR tyrosine kinase inhibitors in EGFR-mutant lung cancer: distinct natural history of patients with tumors harboring the T790M mutation. Clin Cancer Res. 2011 Mar 15;17(6):1616-22. doi: 10.1158/1078-0432.CCR-10-2692. Epub 2010 Dec 6. PMID 21135146
- [Background] Janne PA, Yang JC, Kim DW, Planchard D, Ohe Y, Ramalingam SS, Ahn MJ, Kim SW, Su WC, Horn L, Haggstrom D, Felip E, Kim JH, Frewer P, Cantarini M, Brown KH, Dickinson PA, Ghiorghiu S, Ranson M. AZD9291 in EGFR inhibitor-resistant non-small-cell lung cancer. N Engl J Med. 2015 Apr 30;372(18):1689-99. doi: 10.1056/NEJMoa1411817. PMID 25923549
- [Background] Goss G, Tsai CM, Shepherd FA, Bazhenova L, Lee JS, Chang GC, Crino L, Satouchi M, Chu Q, Hida T, Han JY, Juan O, Dunphy F, Nishio M, Kang JH, Majem M, Mann H, Cantarini M, Ghiorghiu S, Mitsudomi T. Osimertinib for pretreated EGFR Thr790Met-positive advanced non-small-cell lung cancer (AURA2): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1643-1652. doi: 10.1016/S1470-2045(16)30508-3. Epub 2016 Oct 14. PMID 27751847
- [Derived] Mountzios G, Lampaki S, Koliou GA, Vozikis A, Kontogiorgos I, Papantoniou P, Koufaki MI, Res E, Boutis A, Christopoulou A, Pastelli N, Grivas A, Aravantinos G, Lalla E, Oikonomopoulos G, Koumarianou A, Spyratos D, Bafaloukos D, Rigakos G, Papakotoulas P, Fountzilas G, Linardou H. An Observational Study to Assess the Molecular Epidemiology and Direct Medical Costs of Epidermal Growth Factor Receptor (EGFR) Mutations in Patients with Advanced EGFR Mutation-Positive Non-Small Cell Lung Cancer Treated with Afatinib in Real-World Clinical Settings in Greece. Lung Cancer (Auckl). 2021 Aug 30;12:93-102. doi: 10.2147/LCTT.S318007. eCollection 2021. PMID 34512058
- See also: Global Cancer Observatory: Cancer Today; International Agency for Research on Cancer. Estimated Number of New Cases in 2018. — https://gco.iarc.fr/
- See also: World Cancer Research Fund International. Lung cancer statistics — https://www.wcrf.org/dietandcancer/cancer-trends/lung-cancer-statistics